CLINICAL TRIAL: NCT02321020
Title: Sinus Rhythm and Atrial Contractility Recovery After Radiofrequency Maze in Mitral Patients
Brief Title: Follow up of Radiofrequency Maze in Mitral Patients
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Claudia Loardi, MD, Centro Cardiologico Monzino
Other Study IDs: ACFA2
Record Dates: First submitted 2014-12-13; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Radiofrequency maze procedure — Radiofrequency energy was used to create continous endocardial and epicardial lesions mimicking most of the left atrial incisions set as described in the Cox Maze III procedure. In the first 70 patients a monopolar technology was employed (Cardioblate Surgical Ablation Pen, Medtronic Inc, Minneapolis, MN, USA - cooled tip cardioblate pen, power ranging from 25 to 35 W), while in the subset of patients who underwent surgery after July 2005 a bipolar device was used (Cardioblate BP2 Irrigated RF Surgical Ablation System, Medtronic Inc, Minneapolis, MN, USA). The tip of both types of RF probe was irrigated with saline at room temperature at a flow rate of 4-6 ml/min.
Procedure: Transthoracic echocardiography — Contemporary to clinical follow up, all patients were evaluated with 2-dimensional transthoracic echocardiography by the same cardiologist at 3,6,12 and 24 months in order to specifically monitor left atrial contractility presence.

SUMMARY:
The present study aimed at evaluating mid-term results of radiofrequency modified maze procedure in mitral patients in terms of sinus rhythm and atrial contractility restoration

DETAILED DESCRIPTION:
Atrial fibrillation presents with different frequencies in patients affected by structural heart diseases requiring surgery, showing a peak incidence of up to 60-80% in mitral subjects. It causes an increased risk of systemic embolism, cardiac failure development and higher limitations due to dyspnoea and fatigue on exercise. Cox-Maze technique for surgical atrial fibrillation treatment was first used in 1987 and suffered lots of modifications since then. Nowadays, most centers have replaced the "cut and sew" technique by other methods using several power sources to achieve the same target in a much easier way. One of the alternative energy source currently used is radiofrequency ablation which has been demonstrated to be a simple, safe and reproducible procedure with an acceptable success rate in terms of sinus rhythm restoration. However, organized atrial activity (sinus rhythm on surface electrocardiogram) is not always accompanied by an effective mechanical atrial contraction, whose restoration represents one of the original Maze objective. Atrial contraction is effective when A waves are found in tricuspid and/or mitral transvalvular flow using Doppler echocardiography, allowing the patient to fully profit from hemodynamic and clinical advantages of an organized atrial contraction. Predictive factors of atrial contractility recovery and, more widely, of sinus rhythm achievement after modified Maze procedures have been investigated, but, at our knowledge, a parallel deep analysis and comparison of possible determinants of both surgical ablation goals is still lacking. In the present study, the investigators describe mid-term results of concomitant modified radiofrequency Maze in a large homogeneous population of mitral patients, focusing onto common predictors of sinus rhythm and atrial contractility restoring, their time course appearance and interrelation.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by atrial fibrillation undergoing mitral valve surgery

Exclusion Criteria:

* Other cardiac procedures in addition to mitral valve surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by atrial fibrillation undergoing mitral valve surgery
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2002-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sinus rhythm recovery | 5 years
  Early postoperative rhythms were checked in all patients daily by standard 12-channel surface electrocardiogram. Follow up 24 hours Holter monitoring was checked postoperatively at 3,6,12 and 24 months after the intervention and then annually.

SECONDARY OUTCOMES:
Left atrial contractility recovery after maze | 24 months
  All patients were evaluated with 2-dimensional transthoracic echocardiography by the same cardiologist at 3,6,12 and 24 months in order to specifically monitor left atrial contractility presence. Transmitral flow velocity was measured with pulsed Doppler echocardiography, with a sample volume positioned at the level of the mitral tip in the apical four-chamber view and was recorded on a strip chart at a paper speed of 100 mm/s. Peak velocity and the time-velocity integral of the early filling wave (E wave) and of the late filling wave (A wave) were determined. A/E ratio, representing atrial contribution to ventricular diastolic filling, was obtained. Each measurement was obtained as an average of 6 to 8 consecutive beats. Atrial mechanical activity was considered present if an atrial filling (A wave) was detected in late diastole after the electrocardiogram P wave.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Loardi, MD, Principal Investigator — Centro Cardiologico Monzino Milano - Italy